CLINICAL TRIAL: NCT04713436
Title: The Effects of Antibiotic Combinations on Mesenchymal Stem Cells Derived From Apical Papilla
Brief Title: The Effects of Antibiotic Combinations on Stem Cells
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Seçil Çalışkan, Assistant Professor, Eskisehir Osmangazi University
Other Study IDs: 2015-68
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Stem Cells; Anti-Bacterial Agents
MeSH Terms: interventions — Antigens, Differentiation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue samples were obtained from the apex of the extracted third molar teeth of young adult patients aged between 16-22 (N=7).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Triple antibiotic paste(TAP): ciprofloxacin, metronidazole and minocycline
  Interventions: Drug: Differentiation Markers
- Doble antibiotic paste(DAP): ciprofloxacin and metronidazole
  Interventions: Drug: Differentiation Markers
- Modified triple antibiotic paste(mTAP): ciprofloxacin, metronidazole and cefaclor
  Interventions: Drug: Differentiation Markers

INTERVENTIONS:
Drug: Differentiation Markers — Osteocalcin (BGLAP), dentin sialo phosphoprotein (DSPP) and alkaline phosphatase (ALPP) gene expression levels were also evaluated.
  Other Names: Gene expression levels

SUMMARY:
The purpose of this study was to evaluate the indirect effects of antibiotic combinations. SCAP viability, proliferation and apoptosis of the cells were evaluated. Osteocalcin (BGLAP), dentin sialo phosphoprotein (DSPP) and alkaline phosphatase (ALPP) gene expression levels were also evaluated.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the indirect effects of triple (TAP- ciprofloxacin, metronidazole and minocycline), double (DAP- ciprofloxacin and metronidazole) and modified triple antibiotic pastes (mTAP- ciprofloxacin, metronidazole and cefaclor) on mesenchmal stem cells derived from apical papilla (SCAP). SCAP were isolated from the impacted third molar teeth of the young adults. TAP, DAP and mTAP treatment (14-day medication and 28-day medication) were applied on SCAP and viability, proliferation and apoptosis of the cells were evaluated after four weeks. Osteocalcin (BGLAP), dentin sialo phosphoprotein (DSPP) and alkaline phosphatase (ALPP) gene expression levels were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with open apex third molar teeth for extraction indication

Exclusion Criteria:

* Patients with mature apex third molar teeth for extraction indication

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Tissue samples were obtained from the apex of the extracted third molar teeth of young adult patients aged between 16-22 .
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Measurment of Cell Viability and Apoptosis | 1 year
  To evaluate cell viability and apoptosis MuseCell Analyzer Count and Viability kit (Merck Millipore, Taufkirchen, Germany) was used according to the manufacturer's protocol.
Measurment of cell differantiation | 1 year
  To determine gene expression levels, total RNA of SCAP was extracted using the Ambion PureLink RNA mini kit (Invitrogen, US) and the Roche cell RNA Kit (Penzberg, Germany) according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Seçil Çalışkan, Principal Investigator — Eskişehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided